CLINICAL TRIAL: NCT04812964
Title: Modulation of the Intestinal Microbiome in Obesity by a High Protein Diet
Brief Title: Modulation of the Intestinal Microbiome by a High Protein Diet
Acronym: HPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GAST-030-17S
Record Dates: First submitted 2021-03-11; First posted 2021-03-24 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Obesity
Keywords: Obesity; Microbiome; High protein diet
MeSH Terms: conditions — Obesity | interventions — Proteins; Carbohydrates; Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Diet (Active Comparator): Standard protein diet group as control based on 0.5 gram protein per pound of lean body mass with same calories: 15% protein and 55% carbohydrate.
  Interventions: Dietary Supplement: Protein powder supplement, standard dosage based on 0.5 gram protein per pound of subject's lean body mass
- High Protein Diet (Active Comparator): High protein diet group based on 1 gram of protein per pound of lean body mass: 30% protein and 40% carbohydrate.
  Interventions: Dietary Supplement: Protein powder supplement, High Level Protein, based on 1 gram of protein per pound of lean body mass: 25% protein and 45% carbohydrate

INTERVENTIONS:
Dietary Supplement: Protein powder supplement, standard dosage based on 0.5 gram protein per pound of subject's lean body mass — Standard protein diet as control, based on 0.5 gram protein per pound of lean body mass, isocaloric (same number of calories) and consisting of 15% protein and 55% carbohydrate.
  Other Names: Standard Protein Diet
  Arms: Standard Diet
Dietary Supplement: Protein powder supplement, High Level Protein, based on 1 gram of protein per pound of lean body mass: 25% protein and 45% carbohydrate — High level of protein diet, based on 1 gram of protein per pound of subject's lean body mass, isocaloric (same number of calories) and consisting of 30% protein and 40% carbohydrate.
  Other Names: High Protein Diet
  Arms: High Protein Diet

SUMMARY:
The objective of this study is to test and determine whether a high protein diet induces weight loss by modulating the composition and function of the intestinal microbiome in obesity. This will be investigated in a randomized clinical study comparing the effect of isocaloric high and normal protein diets on the intestinal microbiome composition, gene content, and metabolome of obese subjects.

DETAILED DESCRIPTION:
A high protein diet has been shown in preclinical rodent models and clinical trials to be an effective obesity treatment that is associated with greater loss of body weight and fat mass and increased satiety compared to isocaloric standard protein diets. However, the mechanisms of this response have not been fully elucidated. The investigators recently demonstrated in a rodent model that a high protein diet induces shifts in the intestinal microbiome including a bloom of Akkermansia muciniphila, a microbe reported to have an anti-obesity effect. Based on these preliminary studies, the investigators hypothesize that a high protein diet induces alterations in the intestinal microbiome that mediate its clinical efficacy for obesity.

More than three quarters of Veterans are overweight or obese, making obesity a public health problem of tremendous importance to the VA medical system. The results of the proposed study will provide insight into the specific microbes that drive the clinical response to a high protein diet and may identify candidate anti-obesity microbes that could be further developed into novel microbial therapeutics. More broadly, establishing a microbiome-dependent mechanism for the efficacy of a dietary intervention would be a breakthrough in the investigators' understanding of obesity treatment. It would pave the way for larger scale clinical and translational studies investigating the role of the microbiota in other diets and for the development of microbial therapeutics used alone or in combination with dietary intervention to treat obese Veterans.

To investigate the role of the intestinal microbiome in mediating the effect of a high protein diet, the investigators will study 216 overweight and obese Veterans (BMI 27) who will be randomized 1:1 to isocaloric high protein (30%) or normal protein (15%) 1500 calorie diets for 16 weeks utilizing existing clinical infrastructure at the West Los Angeles VA Medical Center established for a recently completed clinical trial of a high protein diet. In Aim 1, the effect of a high protein diet on the composition and function of the intestinal microbiome will be assessed by 16S rRNA sequencing, shotgun metagenomics, and metabolomics. In Aim 2, bioinformatics analysis will be performed to identify fecal microbes, bacterial genes, and metabolites that are associated with weight loss, reduced body fat, decreased hepatic steatosis, altered lipid profiles, reduced hemoglobin A1c, decreased high sensitivity C-reactive protein, increased satiety, and circulating levels of hormones affecting satiety (leptin, ghrelin glucagon, glucagon-like peptide-1, peptide YY).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20 and 60 years of age,
* BMI 27 to 40 kg/m^2,
* non-smoker or stable smoking habits for at least 6 months prior to screening and agreement not to change such habits during the study;
* subjects on non-obesity prescription medication may be included.

Exclusion Criteria:

* Weight change of >3.0 kg in the month prior to screening, weight loss of >10 kg in the 6 months prior to screening,
* calorie restriction diet (<1500 kcal/day) for a period of 4 months or more in the 12 months prior to screening,
* use of any other investigational drug(s) within 8 weeks prior to screening,
* abnormal baseline laboratory parameters (serum creatinine > 1.6 mg/dl; ALT, AST, total bilirubin > 2.0 times the upper limit of normal;
* triglycerides > 500 mg/dl, total cholesterol > 350 mg/dl, TSH outside of normal range),
* consumption of more than 1 alcoholic beverage per day, pregnancy or intention to become pregnant.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Jacobs, MD PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vu JP, Luong L, Parsons WF, Oh S, Sanford D, Gabalski A, Lighton JR, Pisegna JR, Germano PM. Long-Term Intake of a High-Protein Diet Affects Body Phenotype, Metabolism, and Plasma Hormones in Mice. J Nutr. 2017 Dec;147(12):2243-2251. doi: 10.3945/jn.117.257873. Epub 2017 Oct 25. PMID 29070713
- [Background] Dong TS, Luu K, Lagishetty V, Sedighian F, Woo SL, Dreskin BW, Katzka W, Chang C, Zhou Y, Arias-Jayo N, Yang J, Ahdoot A, Li Z, Pisegna JR, Jacobs JP. A High Protein Calorie Restriction Diet Alters the Gut Microbiome in Obesity. Nutrients. 2020 Oct 21;12(10):3221. doi: 10.3390/nu12103221. PMID 33096810
- [Background] Stengel A, Goebel-Stengel M, Wang L, Hu E, Karasawa H, Pisegna JR, Tache Y. High-protein diet selectively reduces fat mass and improves glucose tolerance in Western-type diet-induced obese rats. Am J Physiol Regul Integr Comp Physiol. 2013 Sep 15;305(6):R582-91. doi: 10.1152/ajpregu.00598.2012. Epub 2013 Jul 24. PMID 23883680

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 106 individuals were consented but only 87 completed the first study visit and were considered to have started the study.
Period: Overall Study
Arm/Group | Standard Diet | High Protein Diet
Started | 40 | 47
Completed | 31 | 27
Not Completed | 9 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Diet | High Protein Diet | Total
Number analyzed (Participants) | 40 | 47 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.4) | 56.2 (10.4) | 55.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 29 | 36 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 12 | 17 | 29
  Hispanic | 5 | 13 | 18
  Non-Hispanic White | 20 | 14 | 34
  Asian | 3 | 1 | 4
  Other | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 47 | 87

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss (% Change) in Response to Dietary Intervention Change
Description: The primary objective is to compare weight loss between each of the two diets, a high-protein diet versus a standard protein diet.
Time Frame: Primary outcome of weight loss is measured by subtracting the baseline weight on Day 1 from the weight at the end of the 16 week study period for each subject, and converting to % of baseline weight.
Measure: Mean (Standard Error); unit: percentage weight change from baseline
Arm/Group | Standard Diet | High Protein Diet
Number analyzed (Participants) | 31 | 27
percentage weight change from baseline | -3.83 (0.75) | -3.89 (0.74)

2. Secondary Outcome: Change in Steatosis From Baseline as Measured by Fibroscan in Response to Dietary Intervention
Description: Association of change in fat mass on a high protein diet versus standard protein diet will be measured by Fibroscan (CAP score).
Time Frame: Changes in liver steatosis will be measured at baseline and at the end of the 16 week study period for each subject.
Measure: Mean (Standard Error); unit: dB/m
Arm/Group | Standard Diet | High Protein Diet
Number analyzed (Participants) | 31 | 27
dB/m | -18.3 (13.3) | 3.5 (22.1)

3. Secondary Outcome: Change in Liver Fibrosis From Baseline as Measured by Fibroscan in Response to Dietary Intervention
Description: Association of change in hepatic fibrosis on a high protein diet versus standard protein diet will be measured by Fibroscan elastography.
Time Frame: Changes in liver steatosis will be measured at baseline and at the end of the 16 week study period for each subject.
Measure: Mean (Standard Error); unit: kPa
Arm/Group | Standard Diet | High Protein Diet
Number analyzed (Participants) | 31 | 27
kPa | -1.77 (0.71) | -0.07 (0.57)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Standard Diet | High Protein Diet
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/47
Other Adverse Events (participants affected / at risk) | 0/40 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT04812964/Prot_SAP_000.pdf